CLINICAL TRIAL: NCT05191251
Title: Retrospective Assessment of the Risk of Peripartum Hemorrhage in Pregnant Women : Retrospective Assessment of the Diagnostic Performance of the HEMSTOP Standardized Questionnaire
Status: Completed | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Denis SCHMARTZ, Head, department of Anesthesiology, Brugmann University Hospital
Other Study IDs: CHUB-MAT-HEMSTOP
Record Dates: First submitted 2021-12-29; First posted 2022-01-13 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Peripartum Period; Hemorrhage; HEMSTOP Questionnaire
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Full-term pregnant women with HEMSTOP: Full-term pregnant women who have given birth vaginally or by cesarean section. Patients for whom a HEMSTOP questionnaire could be carried out in prepartum, during the pre-delivery anesthesia consultation.
  Patients who received follow-up during pregnancy as recommended. Age over 18
  Interventions: Diagnostic Test: HEMSTOP questionnaire

INTERVENTIONS:
Diagnostic Test: HEMSTOP questionnaire — A HEMSTOP questionnaire is obtained during the anesthesia consultation.

SUMMARY:
The diagnostic performance of the HEMSTOP (Hematoma, hEmorrhage, Menorrhagia, Surgery, Tooth extraction, Obstetrics, Parents) standardized questionnaire collected during the preoperative anesthesia consultation in order to detect a deficit in hemostasis associated with the risk of hemorrhage in pregnant women will be analyzed. The primary aim of the study is to assess the sensitivity and the specificity of the HEMSTOP questionnaire to identity patients with an abnormal first-line hemostasis test requiring further development by performing second-line hemostasis tests. The second aim of the study is to assess the sensitivity and specificity of the HEMSTOP questionnaire in predicting postpartum hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

Full-term pregnant women who have given birth vaginally or by cesarean section. Patients for whom a HEMSTOP questionnaire could be carried out in prepartum, during the pre-delivery anesthesia consultation.

Patients who received follow-up during pregnancy as recommended. Age over 18

Exclusion Criteria:

Patients age under the age of 18 Patients who did not have follow-up during pregnancy as recommended Patients taking long-term anticoagulants and/or antiaggregants Patients with a language barrier

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Fullterm pregnant women
Study Population: Full-term pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 3588 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity lab tests | 24 hours
  Sensitivity and the specificity of the HEMSTOP questionnaire to identity patients with an abnormal first-line hemostasis test requiring further development by performing second-line hemostasis tests will be calculated.
  Firstline hemostasis tests are aPTT, PT, INR, fibrinogen level and platelet count.

SECONDARY OUTCOMES:
Sensitivity and specificity hemorrhage | 24 hours
  Sensitivity and specificity of the HEMSTOP questionnaire in predicting postpartum hemorrhage will be assessed.
  Postpartum hemorraghe is defined as blood loss greater then 500 mL for vaginal deliveries and greater than 1000 mL for cesarean sections.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bonhomme F, Boehlen F, Clergue F, de Moerloose P. Preoperative hemostatic assessment: a new and simple bleeding questionnaire. Can J Anaesth. 2016 Sep;63(9):1007-15. doi: 10.1007/s12630-016-0688-9. Epub 2016 Jul 1. PMID 27369959
- [Background] Bonhomme F, Ajzenberg N, Schved JF, Molliex S, Samama CM; French Anaesthetic and Intensive Care Committee on Evaluation of Routine Preoperative Testing; French Society of Anaesthesia and Intensive Care. Pre-interventional haemostatic assessment: Guidelines from the French Society of Anaesthesia and Intensive Care. Eur J Anaesthesiol. 2013 Apr;30(4):142-62. doi: 10.1097/EJA.0b013e32835f66cd. PMID 23435255
- [Background] Hawkins JL. Obstetric Hemorrhage. Anesthesiol Clin. 2020 Dec;38(4):839-858. doi: 10.1016/j.anclin.2020.08.010. Epub 2020 Oct 15. PMID 33127031
- [Background] Committee on Practice Bulletins-Obstetrics. Practice Bulletin No. 183: Postpartum Hemorrhage. Obstet Gynecol. 2017 Oct;130(4):e168-e186. doi: 10.1097/AOG.0000000000002351. PMID 28937571
- [Background] Say L, Chou D, Gemmill A, Tuncalp O, Moller AB, Daniels J, Gulmezoglu AM, Temmerman M, Alkema L. Global causes of maternal death: a WHO systematic analysis. Lancet Glob Health. 2014 Jun;2(6):e323-33. doi: 10.1016/S2214-109X(14)70227-X. Epub 2014 May 5. PMID 25103301
- [Background] Al-Zirqi I, Vangen S, Forsen L, Stray-Pedersen B. Prevalence and risk factors of severe obstetric haemorrhage. BJOG. 2008 Sep;115(10):1265-72. doi: 10.1111/j.1471-0528.2008.01859.x. PMID 18715412
- [Background] Butwick A, Lyell D, Goodnough L. How do I manage severe postpartum hemorrhage? Transfusion. 2020 May;60(5):897-907. doi: 10.1111/trf.15794. Epub 2020 Apr 22. PMID 32319687
- [Background] Hoyert DL, Minino AM. Maternal Mortality in the United States: Changes in Coding, Publication, and Data Release, 2018. Natl Vital Stat Rep. 2020 Jan;69(2):1-18. PMID 32510319
- [Background] Eckman MH, Erban JK, Singh SK, Kao GS. Screening for the risk for bleeding or thrombosis. Ann Intern Med. 2003 Feb 4;138(3):W15-24. doi: 10.7326/0003-4819-138-3-200302040-00011-w1. PMID 12558384
- [Derived] Zec T, Schmartz D, Temmerman P, Fils JF, Ickx B, Bonhomme F, Van Der Linden P. Assessment of haemostasis in pregnant women: A retrospective evaluation of the diagnostic performance of the HEMSTOP standardised questionnaire. Eur J Anaesthesiol Intensive Care. 2024 Mar 15;3(2):e0050. doi: 10.1097/EA9.0000000000000050. eCollection 2024 Apr. PMID 39917607